CLINICAL TRIAL: NCT05768087
Title: Escalated Dose Proton Therapy Within the Multimodality Treatment of Glioblastoma Patients - A Phase 1 Proton Dose Finding Trial -
Brief Title: Escalated Dose Proton Therapy Within the Multimodality Treatment of Glioblastoma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-190-22
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Escalated proton therapy (Experimental)
  Interventions: Radiation: Escalated proton therapy

INTERVENTIONS:
Radiation: Escalated proton therapy — According to allocated dose level: level 1-8, 69-90 Gy in 30 fractions of 2.3-3.0 Gy, to a subvolume of the radiation target

SUMMARY:
The goal of this phase 1 dose finding study is to to assess the clinical tolerability and safety of escalated dose proton therapy in glioblastoma patients treated with multimodality treatment, according to treatment volume.

The main questions it aims to answer are:

* what is the maximum tolerated proton dose in glioblastoma patients?
* is the maximum tolerated proton dose in glioblastoma patients dependent on treatment volume?
* what is the recommended phase 2 proton dose in glioblastoma patients?

Patients will be asked to undergo radiotherapy to step-wise escalated doses using proton therapy as part of their multimodality treatment. Patients will be monitored closely for treatment effects.

DETAILED DESCRIPTION:
This is a prospective, single-arm, phase 1 proton dose finding trial, aiming to assess the clinical tolerability and safety of escalated dose proton therapy (PT) in glioblastoma (GBM) patients, according to treatment volume. Radiotherapy will be administered with protons for the entire treatment, escalating the proton fraction-dose with the overall treatment time unchanged. The escalated proton dose will be prescribed to a subvolume of the radiation target. Escalated PT will be employed within the multimodality treatment; surgical procedures and concomitant and adjuvant chemotherapy follow the standard-of-care.

Patients will be subdivided in two groups based on the volume of the radiation target: patients with a CTV2 volume of <200 cc will be placed in group 1 and those with a volume ≥ 200 cc in group 2. Per group, proton dose will be escalated stepwise, which will be guided by a time to event continuous reassessment method (TiTE-CRM) to identify the MTD in this specific combination treatment.

The MTD in this trial is defined as the highest proton dose level at which no more than 30% of the patients develop dose limiting toxicities (DLTs) assessed up to 6 months after the start of PT.

Patient accrual to the main (dose escalation) part of the study ends when the MTD has been identified. If the statistically recommended MTD is declared, an expansion cohort to a total of 6 patients treated at the MTD and 6 patients at the MTD-1 (i.e. 1 dose level below MTD) will be considered. When all patients have been followed for toxicity for at least 1 year after the end of PT (and to a maximum of 2 years), the recommended phase 2 dose (RP2D) will be determined based on the full toxicity profile.

ELIGIBILITY:
Inclusion Criteria (main):

* Newly diagnosed, contrast-enhancing GBM, IDHwt (WHO 2021 classification).
* Maximal safe surgical resection is required; any extent of surgical resection is allowed (including biopsy-only).
* Patient with target volume and location eligible for 60 Gy chemoradiotherapy.
* Minimum distance between GTV and critical OAR (brainstem, chiasm, optic nerves and tracts in case of serviceable vision) of 5 mm on MRI-scan.
* Age ≥ 18 years.
* Karnofsky Performance Status grade of ≥ 70.
* Adequate blood counts as assessed by treating physician.
* Absence of any contraindication to undergo MRI and/or to receive Gadolinium contrast agent.
* Before patient registration, written informed consent must be given according to Good Clinical Practice, and national/local regulations.

Exclusion Criteria:

* All eligibility criteria are formulated as inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | up til 2 years after the end of proton therapy
  CTCAE version 5.0
Dose Limiting Toxicities | up til 6 months after the start of proton therapy
  CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Anouk K Trip, MD PhD, Principal Investigator — Danish Centre for Particle Therapy
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Dept. of Oncology, Aarhus, Central Jutland
  - Danish Centre for Particle Therapy, Aarhus

IPD SHARING:
Plan to Share IPD: No